CLINICAL TRIAL: NCT06866886
Title: Evaluation of the Depth of Sedation in Patients Undergoing Endoscopic Retrograde Cholangio Pancreatography (ERCP) With 4-Channel Electroencephalography (EEG)
Brief Title: EEG-Guided Sedation in ERCP Procedures
Acronym: ERCP-EEG
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayça Özcan, Associate Professor, MD, Ankara City Hospital Bilkent
Other Study IDs: EthicsApproval: E2-24-7125
Record Dates: First submitted 2025-02-24; First posted 2025-03-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Sedation; Sedation Complication; Anesthesia, Intravenous; Monitoring of Depth of Anesthesia; Recovery From Anesthesia
Keywords: patient state index; EEG; ERCP; sedation; PSI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASE GROUP: All patients will undergo routine monitoring, including ECG, blood pressure, SpO₂, respiratory rate, and end-tidal CO₂ measurements. 42 patients receiving EEG-based Patient State Index (PSI) monitoring to optimize sedation depth. PSI electrodes will be applied, and sedation levels will be adjusted accordingly. Oxygen will be administered at 2 L/min via a nasal cannula. Propofol will be used for sedation, with doses adjusted based on patient needs. Any complications that arise and the interventions performed will also be recorded. The procedure duration, total anesthesia duration, total anesthetic dosage, time to awakening from anesthesia (Ramsey Score: 1), and full recovery time (Aldrete Score: 10) will be recorded.
- CONTROL GROUP: All patients will undergo routine monitoring, including ECG, blood pressure, SpO₂, respiratory rate, and end-tidal CO₂ measurements. 42 patients receiving standard clinical sedation monitoring without EEG guidance. Sedation levels will be assessed using the Ramsey Sedation Scale (RSS). Propofol will be used for sedation, with doses adjusted based on patient needs. Oxygen will be administered at 2 L/min via a nasal cannula. Additionally, sedation levels will be evaluated every five minutes using the Ramsey Sedation Scale (RSS). An RSS score of 2-3 will be classified as light sedation, while a score of 4 will indicate deep sedation. Any complications that arise and the interventions performed will also be recorded. The procedure duration, total anesthesia duration, total anesthetic dosage, time to awakening from anesthesia (Ramsey Score: 1), and full recovery time (Aldrete Score: 10) will be recorded.

SUMMARY:
Patients undergoing ERCP have a wide range from patients with poor general condition and septicaemia findings to outpatients who come as day patients without any other additional disease. Rapid deterioration in vital signs may be encountered especially during sedation. In this patient group, it is important to titrate the anaesthetic agent at appropriate doses and to adjust the dose according to the patient.

The aim of the study is to optimise the level of sedation using 4-channel electroencephalography (EEG) in these patients, thus providing balanced anaesthesia and rapid recovery in this already challenging patient group.

DETAILED DESCRIPTION:
Volunteers in the ASA (American Society of Anaesthesiology) I-II-III risk group, aged between 18-65 years, of both sexes, who will undergo ERCP procedure under elective conditions with routine preoperative examination will be included. Before the procedure, the study and all possible risks will be explained to all patients and informed consent will be obtained. Patient's age, weight, ASA value, chronic diseases will be recorded before the procedure. Patients will be divided into two groups. All patients will be routinely monitorised for ECG, non-invasive arterial blood pressure, SpO2, respiratory rate, end-tidal CO2 measurement. These values will be noted at five minute intervals. All patients will receive oxygen at 2 L/min through a nasal cannula. In the case group, in addition to routine monitoring, PSI value measurement will be performed by applying PSI electrodes after wiping the forehead with an alcohol sponge and drying it. All patients will be induced with Propofol at a dose of 1 mg/kg and maintained by infusion at a dose of 50-150 mcg/kg/min according to the patient's need. All procedures will be performed by a single gastroenterologist. In addition, an assessment will be made every five minutes according to the Ramsey Sedation Scale (RSS). An RSS of 2-3 is considered as light sedation and 4 as deep sedation. The duration of the procedure, duration of anaesthesia, total amount of anaesthetic given, time to awakening from anaesthesia (time until Ramsey Score: 1), recovery time (time until Aldrete Score: 10) will be noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III risk score
* Volunteer patients
* Patients aged 18-65 years of both sexes undergoing elective ERCP procedure

Exclusion Criteria:

* Patient reluctance
* Being under 18 years of age
* Being over 65 years of age
* ASA risk score of 4 and above 4
* Pregnant women
* Those with neurological conditions
* Patients with difficult airways
* Obesity (BMI>30)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer patients aged 18-65 years, of both sexes, with ASA I-II-III risk score, undergoing elective ERCP procedure
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Total Anesthetic Consumption | From anesthesia induction to the end of sedation during the ERCP procedure
  The total amount of propofol (mg/kg) administered during the ERCP procedure
Recovery Time from Anesthesia | Assessed at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 minutes post-anesthesia discontinuation, up to 60 minutes.
  The time required for the patient to regain consciousness after anesthesia, defined as the time to reach Aldrete Score of 10
Sedation Depth Maintenance | Sedation depth will be continuously monitored during the procedure and recorded at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes (PSI Score).
  The ability to maintain an optimal sedation level, defined as a Patient State Index (PSI) value around 50, throughout the ERCP procedure.
  Measurement Scale:
  Scale Used: Patient State Index (PSI) - Masimo SedLine Brain Function Monitor Score Range: 0 to 100
  Interpretation:
  0-12: Burst suppression (deep anesthesia) 25-50: Optimal sedation for general anesthesia >50: Light sedation or wakefulness Higher scores indicate lighter sedation, while lower scores indicate deeper sedation.

SECONDARY OUTCOMES:
Hemodynamic Stability | Continuously monitored during the ERCP procedure and recorded at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes.
  Non-Invasive Arterial Blood Pressure (mmHg), including systolic, diastolic, and mean arterial pressure, measured using an automated non-invasive blood pressure monitor to compare intraoperative hemodynamic stability between the EEG-guided sedation group and the standard sedation group.
Hemodynamic Stability | Continuously monitored during the ERCP procedure and recorded at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes.
  Heart Rate (beats per minute), measured using standard ECG monitoring to compare intraoperative heart rate stability between the EEG-guided sedation group and the standard sedation group.
Hemodynamic Stability | Continuously monitored during the ERCP procedure and recorded at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes.
  Oxygen Saturation (SpO₂, %) measured using pulse oximetry to assess intraoperative oxygenation levels in patients undergoing EEG-guided sedation versus standard sedation during the ERCP procedure.
Hemodynamic Stability | Continuously monitored during the ERCP procedure and recorded at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes.
  Respiratory Rate (breaths per minute) measured using continuous respiratory monitoring to assess intraoperative respiratory stability in patients undergoing EEG-guided sedation versus standard sedation during the ERCP procedure.
Hemodynamic Stability | Continuously monitored during the ERCP procedure and recorded at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes.
  End-Tidal CO₂ (mmHg) measured using capnography to assess intraoperative ventilation status and respiratory function in patients undergoing EEG-guided sedation versus standard sedation during the ERCP procedure.
Incidence of Respiratory and Cardiovascular Complications | During the ERCP procedure (intraoperative period)
  The frequency of complications such as hypoxia, apnea, bradycardia, and hypotension
Intervention Rate Due to Sedation-Related Instability | During the ERCP procedure (intraoperative period)
  The need for additional interventions such as airway support, fluid therapy, vasopressors, or increased oxygen administration due to sedation-related complications
Time to Awakening from Anesthesia | Assessed at 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 minutes post-anesthesia discontinuation, up to 60 minutes.
  The time taken for the patient to regain consciousness, defined as the time to reach Ramsey Sedation Score (RSS) of 1.
  Scale Used: Ramsey Sedation Scale (RSS) Score Range: 1 to 6
  Interpretation:
  1: Patient is awake, anxious, and agitated 2-3: Light sedation (responsive to verbal commands) 4: Deep sedation (responsive to light stimuli) 5-6: Unresponsive to stimuli (very deep sedation) Higher scores indicate deeper sedation, while lower scores indicate increased wakefulness.
Total Procedure Duration | From the start to the completion of the ERCP procedure
  The overall time taken to complete the ERCP procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Özcan, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No